CLINICAL TRIAL: NCT00454506
Title: Prospective Evaluation of the Clinical and Economic Outcomes of Total Joint Replacement: HSS Hip Arthroplasty Cohort
Brief Title: Hospital for Special Surgery Hip Arthroplasty Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2015-092
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Total joint replacements are some of the most successful medical devices developed over the last fifty years. They enable millions of people to remain ambulatory and pain free, with minimal risk. In 2002, over 200,000 total hip replacements, 350,000 total knee replacements, and 25,000 total or partial shoulder replacements were performed in the United States (HCUP data). Future use will likely be even higher: it is estimated that by the year 2020, the population 65 and over in developed countries will increase by 71%. Existing studies do not provide adequate prospective data to evaluate long-term outcomes. Most health related quality of life studies in THA and TKA only report data up to twelve months post-operatively. In addition, most large studies of TKA and THA have been performed in Medicare patients. While these databases are important in providing population based data, Medicare studies do not permit any direct patient contact, and provide no information on patients under 65.

Existing studies have also investigated predictors of patient outcome at one and two years after joint arthroplasty. However, very little is known about predictors of prosthesis failure, and there are no validated clinical indicators for choosing one prosthesis model over another. Once a device is FDA approved, there is very little motivation on the part of the developer to perform complete post-marketing research, despite the importance of these data to the public health. Most existent studies are not powered to compare differences between models.

The purpose of this study is to establish a prospective cohort of HSS total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing total knee arthroplasty at HSS
* Pregnant women are eligible for the registry as this is a non-interventional study which only involves filling out questionnaires.

Exclusion Criteria:

* No other exclusion criteria;this is a non-interventional study which only involves filling out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be asking all patients undergoing a total hip arthroplasty to participate.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Sculco, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: CERTs tools and resources — http://certs.hhs.gov